CLINICAL TRIAL: NCT01029964
Title: A Three-year Behavioral Treatment of Obese Children: the Effect of Age on Change in BMI SDS and Dropout Rate
Brief Title: A Three-year Behavioral Treatment of Obese Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Claude Marcus Professor, Karolinska Institutet
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BORIS
Record Dates: First submitted 2009-12-09; First posted 2009-12-10 (Estimated); Last update posted 2009-12-10 (Estimated); Status verified 1997-01

CONDITIONS: Childhood Obesity
Keywords: Childhood obesity; Age-dependent; Long-term treatment; BMI SDS; Dropouts
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 6-9 years (Active Comparator): Age at start of treatment
  Interventions: Behavioral: Individually and in groups
- 10-13 years (Active Comparator): Age at start of treatment
  Interventions: Behavioral: Individually and in groups
- 14-16 years (Active Comparator): Age at start of treatment
  Interventions: Behavioral: Individually and in groups
- Control 6-9 years (No Intervention): Untreated control group

INTERVENTIONS:
Behavioral: Individually and in groups — During three year in a clinical setting.
  Arms: 10-13 years; 14-16 years; 6-9 years

SUMMARY:
The prevalence of overweight and obesity among children and adolescents has reached epidemic proportions worldwide. Among Swedish 10-year old children 15-20% are overweight and 3-5% are obese. The probability that an obese child becomes an obese adult is very high. This chronic disease requires lifetime treatment. The standard treatment of childhood obesity involves behavioural interventions focused on eating habits and physical activity. Studies often include small study samples, the absence of control groups and short treatments times. Several long-term follow-up studies of shorter interventions are available. The results from these studies are disappointing since the number of children who are "cured" i.e., have become non-obese is low. Thus, effective treatments are currently lacking.The National Childhood Obesity Center treats children in a University hospital setting. The children are enrolled from the catchment areas of the hospital as well as the rest of Sweden. Treatment alternatives include behavioural treatment (individual and group), low and very low calorie diet, pharmacological and surgical treatment. Patients treated with surgical and pharmacological methods safety is ensured using these treatments exclusively in controlled studies. The clinic was the first in Sweden with this wide range of treatment options.

BORIS is a national health care quality register for childhood obesity, supervised by the Swedish Association of Local Authority and Regions.

DETAILED DESCRIPTION:
The primary aim of this study was to compare treatment effects (changes in BMI SDS) during the first three years of behavioral treatment in relation to age at start of treatment. The secondary aim was to evaluate specific factors of importance (gender, heredity, parental weight status, socioeconomic factors and age at obesity onset) for treatment effects. The third aim was to investigate factors correlated to drop out.

This is a longitudinal study of all patients referred to National Childhood Obesity Center between January 1997 and December 2004. Only patients with behavioral treatment were included. Patients with other treatments (VLCD/LCD, drugs and surgery) and other diagnoses (syndromes, craniopharyngioma, Mb Down, myelomeningocele, various types of mental and psychological disorders) and children <6 and >17 year at inclusion were excluded. The remaining children were divided into three age groups of obese children depending of age at onset of obesity treatment (6-9, 10-13 and 14-16year). All patient data were registered in the BORIS nationwide childhood obesity database.

ELIGIBILITY:
Inclusion Criteria:

* All children treated with behavioral treatment at the National childhood obesity center Stockholm between january 1998 - december 2004.
* Classified as obese by using the Tim Cole standard.

Exclusion Criteria:

* Children with obesity together with other diagnosis
* Children with other treatment like pharmacological, low calorie diets and surgery

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1000 (Actual)
Dates: Start 1997-01; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Measured as change in BMI SDS. | Three years behavioral treatment

CONTACTS AND LOCATIONS:
Overall Officials: Claude Marcus, Professor, Principal Investigator — 1National Childhood Obesity Center, Children´s Hospital, Karolinska University Hospital, Karolinska Institutet, Dept. of Clinical Science, Intervention and Technology (CLINTEC), Division of Pediatrics, Stockholm, Sweden
Locations (1):
- Karolinska University Hospital, Karolinska Institutet, Dept. of Clinical Science, Intervention and Technology (CLINTEC), Division of Pediatrics, Stockholm, Huddinge, Sweden

REFERENCES:
- [Derived] Danielsson P, Svensson V, Kowalski J, Nyberg G, Ekblom O, Marcus C. Importance of age for 3-year continuous behavioral obesity treatment success and dropout rate. Obes Facts. 2012;5(1):34-44. doi: 10.1159/000336060. Epub 2012 Mar 2. PMID 22433615